CLINICAL TRIAL: NCT02736825
Title: Non-Inferiority Study of the Safety and Efficacy of Ultherapy® Using Standard Versus Simulines Transducers at a Reduced Energy Level for Patient Comfort
Brief Title: Simulines Non-Inferiority Pivotal Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study data to date show the required primary study endpoint will not be met.
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULT-146
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2018-01

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A, Ulthera System with standard transducers (Active Comparator): Subjects randomized to Group A will receive an Ultherapy® treatment to the lower face and neck with a total minimum pulse count of 672 pulses (+5%) at the 4.5mm and 3.0mm depths using standard transducers. Energy levels for each transducer will be set to EL2:
  * Deep-See (DS) 4-4.5 at 0.9 Joules (J) with pitch of 1.5mm and 17 Thermal Coagulation Points (TCP)s per line
  * DS 7-3.0 at 0.30J with pitch of 1.1mm and 23 TCPs per line
  Interventions: Device: Ulthera System with standard transducer
- Group B, Ulthera System with prototype 2 simulines transducers (Experimental): Subjects randomized to Group B will receive a Ultherapy® treatment with a total minimum pulse count of 336 pulses (+5%) using the prototype 2 simulines transducers at the 4.5mm and 3.0mm depths. Energy levels for each transducer will be set to EL2:
  * Deep-See 4-4.5 Simulines (DS 4-4.5S) at 1.23J with pitch of 1.5mm and 17 TCPs per line
  * DS 4-3.0S at 0.88J with pitch of 1.3mm and 20 TCPs per line
  Interventions: Device: Ulthera System with prototype 2 simulines transducer

INTERVENTIONS:
Device: Ulthera System with standard transducer — Focused ultrasound energy delivered below the surface of the skin using commercially available transducer to deliver one line of treatment at a time
  Other Names: Ultherapy
  Arms: Group A, Ulthera System with standard transducers
Device: Ulthera System with prototype 2 simulines transducer — Focused ultrasound energy delivered below the surface of the skin using new transducer to deliver two lines of treatment simultaneously
  Other Names: Ultherapy
  Arms: Group B, Ulthera System with prototype 2 simulines transducers

SUMMARY:
Up to 260 subjects presenting with skin laxity on the face and neck will be randomized to one of two treatment groups. Subjects meeting all entrance criteria will receive study treatment, then complete two post treatment phone contacts and follow-up study visits at 90, 180 and 365 days post treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit for qualitative and quantitative assessments of efficacy.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blinded, multi-center, parallel arm, non-inferiority, pivotal clinical trial to demonstrate the efficacy of the Ultherapy treatment with prototype 2 simulines transducers (4-3.0 Smm and 4-4.5 Smm) at energy level (EL) 2 is non-inferior to treatment with standard transducers (7-3.0 mm and 4-4.5mm) at EL 2 for lifting the lower face and neck and to demonstrate the safety of treatment with prototype 2 simulines transducers is similar to treatment with standard transducers.

Changes from baseline in quantitative measures of neck and submental lift will be assessed at study follow-up visits. Global Aesthetic Improvement Scale scores, Merz Jawline Grading Scale scores, 3D volumetric changes from baseline to post treatment, patient satisfaction and patient-reported improvement will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 70 years.
* Subject in good health.
* Body Mass Index (BMI) of ≤30.
* Skin laxity in the area(s) to be treated as determined by trained physician assessors.
* Willingness to avoid excessive or prolonged exposure to sunlight, tanning booths, sun lamps, or ultraviolet (UV) light sources.
* Willingness to apply study provided sunscreen (Neocutis Micro-Day Rejuvenating Cream) daily until study exit to help limit sun exposure.
* Willingness to avoid or periodically stop use of Sunless Tanners (washout period of two weeks prior to each study visit is required).
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period
* Willingness to avoid non-emergent dental procedures in the 3 weeks prior to/ post treatment.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, intrauterine device (IUD), surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

  a. Postmenopausal for at least 12 months prior to study; b. Without a uterus and/or both ovaries; or c. Bilateral tubal ligation at least six months prior to study enrollment.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other non-steroidal anti-inflammatory drug (NSAID) prior to study treatment and chronic use during the entire post-treatment study period. Washout period, if chronic user, for 4 weeks prior to the study treatment. After study treatment is completed, limited acute NSAID use, i.e., a maximum of 2-3 doses in any 2 week period, is allowed if needed.
* Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* History of Bell's Palsy.
* History of chronic or frequently recurring episodic (recurrent episode in past 12 months) autoimmune diseases such as Multiple Sclerosis, Crohn's Disease, Psoriasis, Myasthenia Gravis, Lambert-Eaton Syndrome that has required immune suppressant therapy (such as biologic drug or corticosteroid treatment).
* Palpable thyroid lesion, lymphadenopathy, or other pathological changes within the treatment area.
* History of skin cancer in the areas to be treated, basal cell nevus syndrome, or jaw cysts.
* Known allergy or sensitivity to Ibuprofen.
* Severe solar elastosis.
* BMI > 30.
* Significant changes in weight (e.g. more than 5 pounds) over the past 6 months or anticipated significant changes in weight or diet over the course of the study.
* Pregnant within the past year.
* Excessive subcutaneous fat in the area(s) to be treated.
* Excessive skin laxity in the area(s) to be treated as determined by trained physician assessors.
* Significant scarring in the area(s) to be treated that would interfere with assessing results.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included).
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within two weeks prior to study participation or during the study.
* Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
* History of chronic drug or alcohol abuse.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
* History of the following cosmetic treatments in the area(s) to be treated:

  1. Any energy based device (radio-frequency (RF), micro-focused ultrasound (MFU), etc.) procedure for skin tightening within the past year;
  2. Injectable filler of any type within the past:

  i. 12 months for Hyaluronic acid fillers (e.g. Restylane)

ii. 12 months for Ca Hydroxylapatite fillers (e.g. Radiesse)

iii. 24 months for Long Lasting Hyaluronic acid (e.g. Voluma) and Poly-L-Lactic acid fillers (e.g. Sculptra)

iv. Ever for permanent fillers (e.g. Silicone, ArteFill)

c. Neurotoxins within the past six months (neuromodulators are allowed in the glabella and forehead, not allowed in the temples, crow's fee or anywhere below the lateral canthus);

d. Fractional and fully ablative resurfacing laser treatment within the past two years;

e. Nonablative, rejuvenative laser or light treatment within the past six months;

f. Surgical dermabrasion or deep facial peels within the past two years;

g. Facelifts, neck surgery (e.g. thyroid, neck lifts, neck liposuction, etc.) within the past two years;

h. Micro needling within the past year;

i. Kybella, Coolsculpting, or Mesotherapy within the past two years; or

j. Any history of contour threads.

* History (in the prior year) or current use of the following prescription medications:

  1. Accutane or other systemic retinoids within the past six months;
  2. Initiation of topical retinoids within the past 6 months or throughout the course of the study;
  3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix);
  4. Systemic steroids including prednisone;
  5. Dermal regulators of collagen;
  6. Initiation of bioidentical hormones or human growth hormone (HGH) within the past 6 months or throughout the course of the study; or
  7. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Ulthera, Inc
Locations (8):
- United States (8):
  - Clinical Testing of Beverly Hills, Beverly Hills, California
  - Roseville Facial Plastic Surgery, Roseville, California
  - Laser and Skin Surgery Center, Sacramento, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, San Diego, California
  - AboutSkin Dermatology, Greenwood Village, Colorado
  - Maryland Laser Skin and Vein Dermatology, Cockeysville, Maryland
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 sites in the United States.
Pre-assignment Details: A total of 262 participants were screened, enrolled, and treated in the study. Of these, 240 participants completed the 180-days evaluation. The study was terminated at 180 days.
Groups:
- Group A: Participants received single Ultherapy treatment to the lower face and neck with a total minimum pulse count of 672 pulses (+5 percent [%]) at the 4.5 millimeter (mm) and 3.0 mm depths at EL 2, using standard transducers DeepSEE (DS) 4-4.5 at 0.9 joules (J) with pitch of 1.5 mm and 17 thermal coagulation points (TCPs) per line and DS 7-3.0 at 0.30 J with pitch of 1.1 mm and 23 TCPs per line.
- Group B: Participants received single Ultherapy treatment to the lower face and neck with a total minimum pulse count of 336 pulses (+5%) at the 4.5 mm and 3.0 mm depths at EL 2 using prototype 2 simulines transducers DS 4-4.5S at 1.23 J with pitch of 1.5 mm and 17 TCPs per line and DS 4-3.0S at 0.88 J with pitch of 1.3 mm and 20 TCPs per line.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 127 | 135
Completed | 117 | 123
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 10 | 11
Not completed — Early Termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was the subset of all participants who were exposed to study treatment at least once.
Groups:
- Group A: Participants received single Ultherapy treatment to the lower face and neck with a total minimum pulse count of 672 pulses (+5 %) at the 4.5 mm and 3.0 mm depths at EL 2, using standard transducers DS 4-4.5 at 0.9 J with pitch of 1.5 mm and 17 TCPs per line and DS 7-3.0 at 0.30 J with pitch of 1.1 mm and 23 TCPs per line.
- Group B: Participants received single comparable treatment with a total minimum pulse count of 336 pulses (+5%) at the 4.5 mm and 3.0 mm depths at EL 2 using prototype 2 simulines transducer DS 4-4.5 at 1.23 J with pitch of 1.5 mm and 17 TCPs per line and DS 4-3.0 S at 0.88 J with pitch of 1.3 mm and 20 TCPs per line.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 127 | 135 | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (7.3) | 52.6 (8.0) | 53.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 129 | 245
  Male | 11 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Black/African American | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  White | 123 | 127 | 250
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127 | 135 | 262
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 65.5 (3.0) | 65.3 (3.0) | 65.4 (3.0)
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 145.1 (23.0) | 142.1 (22.3) | 143.6 (22.6)
Body mass index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 23.7 (2.8) | 23.4 (2.8) | 23.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Greater Than or Equal to (>=) 20 mm^2 Reduction in Submental Area at Day 90
Description: Participant response was defined as >=20 mm^2 reduction in 2D submental area from baseline. Submandibular and Submental quantitative measurements were calculated comparing participants using prototype 2 simulines versus standard transducers. The standard 2D photographic images were obtained. Utilizing the lateral profile view of pre-and 90-day post treatment photos of each participant, quantitative results were calculated by using 5 evenly spaced points on the neck. Area was calculated between each of the 5 points and then sum of the 5 calculations was the total area of the region of interest. The delta area between the pre-and post-treatment area of the chin and neck determined the amount of tissue lift in the area.
Time Frame: Day 90
Population: The intent-to-treat (ITT) population consisted of all participants in the SES for whom the primary efficacy variable was available.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 126 | 132
Participants | 64 | 50
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Non-Inferiority — Non-inferiority margin of 15% between two independent percentages using the z-test with unpooled variance; p = 0.3670, Z-test

2. Secondary Outcome: Number of Participants Who Achieved >=20 mm^2 Reduction in Submental Area at Day 180
Description: Participant response was defined as >=20 mm^2 reduction in 2D submental area from baseline. Submandibular and Submental quantitative measurements were calculated comparing participants using prototype 2 simulines versus standard transducers. The standard 2D photographic images were obtained. Utilizing the lateral profile view of pre-and 180-day post treatment photos of each participant, quantitative results were calculated by using 5 evenly spaced points on the neck. Area was calculated between each of the 5 points and then sum of the 5 calculations was the total area of the region of interest. The delta area between the pre-and post-treatment area of the chin and neck determined the amount of tissue lift in the area.
Time Frame: Day 180
Population: No data was collected because the study was terminated at 180 days.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Who Achieved >=20 mm^2 Reduction in Submental Area at Day 365
Description: as for outcome 2
Time Frame: Day 365
Population: No data was collected because the study was terminated at 180 days.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants Who Showed Improvement in Overall Lifting and Tightening of Skin at Day 90
Description: Improvement was determined by qualitative assessment of photographs by a masked physician.
Time Frame: Day 90
Population: The ITT population consisted of all participants in the SES for whom the primary efficacy variable was available.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 126 | 132
Participants | 67 | 51

5. Secondary Outcome: Number of Participants Who Showed Improvement in Overall Lifting and Tightening of Skin at Day 180
Description: Improvement was determined by qualitative assessment of photographs by a masked physician.
Time Frame: Day 180
Population: The ITT population consisted of all participants in the SES for whom the primary efficacy variable was available. Participants who were evaluable for this measure at given time period were included.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 117 | 123
Participants | 55 | 54

6. Secondary Outcome: Number of Participants Who Showed Improvement in Overall Lifting and Tightening of Skin at Day 365
Description: Improvement was determined by qualitative assessment of photographs by a masked physician.
Time Frame: Day 365
Population: No data was collected because the study was terminated at 180 days.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in Volume as Assessed by Quantificare 3 D Imaging System at Day 90
Description: Additional images were obtained using a 3D digital photo system. QuantifiCare 3D imaging was used to assess the volumetric changes. Four views (Face, UnderRight, UnderLeft, and Neck) were compared for each participant.
Time Frame: Day 90
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 7 | 8
Percent change | -0.8 (4.3) | -4.1 (5.0)

8. Secondary Outcome: Percent Change From Baseline in Volume as Assessed by Quantificare 3D Imaging System at Day 180
Description: as for outcome 7
Time Frame: Day 180
Population: The ITT population consisted of all participants in the SES for whom the primary efficacy variable was available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 7 | 8
Percent change | -4.7 (5.6) | 0.5 (4.5)

9. Secondary Outcome: Percent Change From Baseline in Volume as Assessed by Quantificare 3D Imaging System at Day 365
Description: as for outcome 7
Time Frame: Day 365
Population: No data was collected because the study was terminated at 180 days.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Some Level of Improvement and Satisfaction on Day 90
Description: Participants completed a patient satisfaction questionnaire (PSQ) at the 90-day visit. The PSQ has 5 improvement and satisfaction categories ranging from "worse" to "much improved" and "dissatisfied' to "very satisfied".
Time Frame: Day 90
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 125 | 132
Participants
  Much improved | 23 | 10
  Improved | 30 | 35
  A little improved | 48 | 49
  No change | 21 | 36
  Worse | 3 | 2
  Very satisfied | 21 | 10
  Satisfied | 40 | 40
  Slightly satisfied | 28 | 37
  Neither satisfied or dissatisfied | 26 | 37
  Dissatisfied | 10 | 8

11. Secondary Outcome: Mean Treatment Times
Description: Mean treatment time was based on a comparison of average time to complete treatment using each transducer type. The time to complete the study treatment for each group was recorded on the system treatment logs as treatment start time (time treatment started on the Ulthera system) and stop time (time treatment ended on the Ulthera system).
Time Frame: Baseline
Population: The SES was the subset of all participants who were exposed to study treatment at least once.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group A | Group B
Number analyzed (Participants) | 127 | 135
Minutes | 55.6 (15.2) | 33.1 (11.4)

12. Secondary Outcome: Mean Pain Scores to Assess Participant's Treatment Related Comfort Level Based on Numeric Rating Scale (NRS)
Description: Participant's treatment-related pain scores were obtained using a validated 11-point NRS with 0: no pain; 5: moderate pain; and 10: worst possible pain. Pain scores were obtained following each region treated (submandibular/submental and cheeks) and for each transducer used during treatment. Average pain score was calculated for each arm by adding all the scores of all participants in each arm to obtain the mean NRS score.
Time Frame: Baseline
Population: The SES was the subset of all participants who were exposed to study treatment at least once.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 127 | 135
Score on a scale
  4.5 mm Depth | 5.5 (2.1) | 4.6 (2.0)
  3.0 mm Depth | 3.1 (1.8) | 4.6 (2.1)

13. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by Subject Global Aesthetic Improvement Scale (SGAIS) at Day 90
Description: Overall aesthetic improvement was assessed by participants using SGAIS. Each participant completed a SGAIS. The SGAIS was 5-point scale (1-5), where: 1 (very much improved); 2 (much improved); 3 (improved); 4 (no change); 5 (worse).
Time Frame: Day 90
Population: The ITT population consisted of all participants in SES for whom primary efficacy variable was available.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 126 | 132
Participants
  Very much improved | 12 | 3
  Much improved | 18 | 13
  Improved | 55 | 73
  No change | 37 | 41
  Worse | 4 | 2

14. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by SGAIS at Day 180
Description: as for outcome 13
Time Frame: Day 180
Population: The ITT population consisted of all participants in SES for whom primary efficacy variable was available. Participants who were evaluable for this measure at given time period were included.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 118 | 127
Participants
  Very much improved | 9 | 10
  Much improved | 18 | 18
  Improved | 53 | 62
  No change | 36 | 34
  Worse | 2 | 3

15. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by SGAIS at Day 365
Description: as for outcome 13
Time Frame: Day 365
Population: No data was collected because the study was terminated at 180 days.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by Clinician Global Aesthetic Improvement Scale (CGAIS) at Day 90
Description: Overall aesthetic improvement was assessed by the clinician using a CGAIS. The CGAIS was 5-point scale (1-5), where: 1 (very much improved); 2 (much improved); 3 (improved); 4 (no change); 5 (worse).
Time Frame: Day 90
Population: The ITT population consisted of all participants in SES for whom primary efficacy variable was available.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 126 | 132
Participants
  Very much improved | 10 | 8
  Much improved | 33 | 34
  Improved | 63 | 65
  No change | 20 | 24
  Worse | 0 | 1

17. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by CGAIS at Day 180
Description: as for outcome 16
Time Frame: Day 180
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 118 | 127
Participants
  Very much improved | 5 | 11
  Much improved | 32 | 20
  Improved | 57 | 68
  No change | 24 | 28
  Worse | 0 | 0

18. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by CGAIS at Day 365
Description: as for outcome 16
Time Frame: Day 365
Population: No data was collected because the study was terminated at 180 days.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 180 days
Description: The investigator asked the participant for adverse events systematically at each visit.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/135
Other Adverse Events (participants affected / at risk) | 24/127 | 14/135
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=127) | Group B (N=135)
Bruising/Ecchymosis (General disorders) | 4 | 3
Edema (General disorders) | 12 | 4
Tenderness/Soreness/Pain/ Sensitivity to Touch (General disorders) | 15 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT02736825/Prot_SAP_000.pdf